CLINICAL TRIAL: NCT01071161
Title: Phase III (c) The Effect of Azithromycin in Patients With COPD and Chronic Productive Cough
Brief Title: The Effect of Azithromycin in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Productive Cough
Acronym: CACTUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL19886.075.08
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Cough; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: chronic cough; COPD; Azithromycin; Zithromax; LCQ
MeSH Terms: conditions — Cough; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Chronic Cough | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Experimental)
  Interventions: Drug: azithromycin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: azithromycin — azithromycin, tablets, during 12 weeks, three times a week, 250mg
  Other Names: Zithromax
  Arms: Azithromycin
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of azithromycin to produce a significant change in the cough-related health status, measured with the Dutch version of the Leicester Cough Questionnaire in patiënts with COPD gold classification 2-4 and chronic productive coughing.

DETAILED DESCRIPTION:
This study is a prospective double-centre, double blind randomised trial. Patients > 40 years of age, referred to our outpatient clinic with chronic cough and sputum production due to COPD will be recruited after informed consent is obtained.

Consenting patients will be randomises to a 12-week treatment with 250 mg azithromycin three times a week or placebo.

Before randomisation all patients have to fill in the SF 36 , SGRQ and the Dutch version of the Leicester Cough Questionnaire (LCQ) for assessment of the baseline quality of life and the disease specific quality of life.

The LCQ questionnaires will be performed at the beginning and every 3 weeks afterwards until 18 weeks, except the second LCQ which will be filled in after 2 weeks. Scores from this questionnaire will be used to calculate the 2-week repeatability. The SF 36 and SGRQ will be performed at the start of the study and after 12 weeks. Adverse events will be recorded during the whole treatment period. After 2 and 12 weeks a Global Rating of Change will be performed. This questionnaire will be used to validate the LCQ in COPD patients.

Randomisation will take place using a computer allocation program (BAMI-computer)

Azithromycin and placebo will be provided by Teva Pharmaceuticals. Placebo and azithromycin will be identical in appearance and packaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years of age, in our outpatient clinic with chronic cough and COPD (gold2-4)
* Chronic cough is defined as a cough > 12 weeks duration, at least 12 weeks a year in 2 subsequent years.
* Analysed for bronchiectasis prior to participation by CT-thorax.

Exclusion Criteria:

* Prior history of asthma
* Use of i.v. or oral corticosteroids and or antibiotics for an exacerbation 3 weeks before inclusion
* Patients suffering from other relevant lung diseases.
* Clinically relevant abnormal laboratory values suggesting an unknown disease requiring further clinical evaluation.
* Liver disease, (ALAT and/or ASAT levels two or more times the upper limit of normal).
* Pregnancy or lactation.
* Use of macrolides the last 6 weeks prior to inclusion.
* Allergy or intolerance to macrolides.
* Other research medication started 2 months prior to inclusion.
* Prior randomisation in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mean change in the Leicester Cough Questionnaire (LCQ) scores. | 2 years

SECONDARY OUTCOMES:
Mean change in the SF 36 and SGRQ scores. | 2 years
Change in lung function, (FEV1 (L) and FVC (L)). | 2 years
Number of exacerbations. | 2 years
Adverse reactions. | 2 years
Laboratory values: CRP, ASAT, ALAT | 2 years
Sputum analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan W van den Berg, MD, Study Director — Department of Pulmonology
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Derived] Berkhof FF, Doornewaard-ten Hertog NE, Uil SM, Kerstjens HA, van den Berg JW. Azithromycin and cough-specific health status in patients with chronic obstructive pulmonary disease and chronic cough: a randomised controlled trial. Respir Res. 2013 Nov 14;14(1):125. doi: 10.1186/1465-9921-14-125. PMID 24229360
- [Derived] Berkhof FF, Boom LN, ten Hertog NE, Uil SM, Kerstjens HA, van den Berg JW. The validity and precision of the Leicester Cough Questionnaire in COPD patients with chronic cough. Health Qual Life Outcomes. 2012 Jan 9;10:4. doi: 10.1186/1477-7525-10-4. PMID 22230731